CLINICAL TRIAL: NCT00503568
Title: Novel Tumor Vaccine gp96-Ig Fusion Protein in Advanced (Stage IIIB), Relapsed or Metastatic (Stage IV) Non-Small Cell Lung Cancer (NSCLC) Patients Who Have Failed First Line Chemotherapy
Brief Title: Vaccine Therapy in Treating Patients With Stage III, Stage IV, or Relapsed Non-Small Cell Lung Cancer Treated With First-Line Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020225; SCCC-2002041 (Other: UM/Sylvester Comprehensive Cancer Canter); WIRB-20050969 (Other: Western IRB); NCT00247065 (obsolete NCT alias)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DS-1: gp96-ig Dose Schedule 1 (Experimental): Dose Schedule 1 (DS-1): Ad100-gp96Ig-HLA A1 Vaccine 4x10^7 cells bi-weekly, maximum 9 vaccines/patient;
  Interventions: Biological: Ad100-gp96Ig-HLA A1
- DS-2: gp96-ig Dose Schedule 3 (Experimental): Dose Schedule 2 (DS-2): Ad100-gp96Ig-HLA A1 Vaccine 2X10^7 cells weekly, maximum 18 vaccines/patient;
  Interventions: Biological: Ad100-gp96Ig-HLA A1
- DS-3: gp96-ig Dose Schedule 3 (Experimental): Dose Schedule 3 (DS-3): Ad100-gp96Ig-HLA A1 Vaccine 1x10^7 cells twice weekly, maximum 36 vaccines/patient
  Interventions: Biological: Ad100-gp96Ig-HLA A1

INTERVENTIONS:
Biological: Ad100-gp96Ig-HLA A1 — Dose Schedule 1 (DS-1): 4x10^7 cells bi-weekly, maximum 9 vaccines/patient; Dose Schedule 2 (DS-2): 2X10^7 cells weekly, maximum 18 vaccines/patient; Dose Schedule 3 (DS-3): 1x10^7 cells twice weekly, maximum 36 vaccines/patient
  Other Names: gp96-vaccine; gp96-Ig and HLA A1 transfected Non-Small Cell Lung Cancer cell line

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells may help the body build an effective immune response to kill non-small cell lung cancer cells.

PURPOSE: This phase I trial is studying the effects of gp96-Ig vaccine therapy in treating patients with stage III, stage IV, or relapsed non-small cell lung cancer treated with first-line chemotherapy.

DETAILED DESCRIPTION:
Overall Goals:

- to evaluate the safety and induction of anti-tumor immunity by administration of an immunogenic human tumor cell vaccine, and assess immune response in relation to clinical outcome.

Primary Aim:

- to evaluate the safety of administering a heat shock protein gp96-Ig-secreting allogeneic tumor cell-vaccine (gp96-Ig vaccine) in patients with advanced NSCLC.

Secondary Aims:

* to study the immune response to vaccination,
* to monitor clinical responses and
* to recommend a dose-schedule combination for further testing in an initial Phase II trial of vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed NSCLC (squamous, adeno-, large cell anaplastic, bronchoalveolar, and non-small cell carcinoma NOS): stage IIIB with malignant pleural effusion, stage IV, or recurrent disease.
* At least one site of bi-dimensionally measurable disease.
* Metastasis if present and treated must be stable by CT scan or MRI for at least 8 weeks.
* Patient must have received and failed at least one line of chemotherapy.
* Age >= 18 years.
* ECOG performance status 0-2.
* Life expectancy >= 3 months.
* Laboratory parameters:

  * Hemoglobin levels >= 10.0 (transfusions allowed if necessary).
  * ANC >= 1,500.
  * Platelets >= 100k.
  * Creatinine clearance >= 50 ml/min.
  * Total and direct bilirubin: < 2.5 X upper institution limit for normal.
  * Liver function tests: AST, ALT, and AlkP < 2.5 X upper institution limit for normal.
* Signed informed consent.
* Autopsy consent - although not a requirement for study entry, patients who consent to participate in study will be made aware of the critical importance of a post-mortem examination in the event of the patient's death after receiving therapy with this experimental vaccine. Therefore, pre-treatment written agreement to autopsy will be sought from the patient, or verbal agreement to autopsy will be sought in the presence of the next of kin or other family members.

Exclusion Criteria

* Active or symptomatic cardiac disease such as congestive heart failure, angina pectoris or recent myocardial infarction. Patients with history of these conditions who are stable taking cardiac medications will also be excluded.
* Pregnant or lactating women (negative test for pregnancy is required of women of childbearing potential).
* Known HIV infection.
* Uncontrolled or untreated brain or spinal cord metastases.
* Active infection.
* Concomitant steroid or other immunosuppressive therapy.
* Other active malignancies present within the past three years, except for basal and/or squamous cell carcinoma(s) or in situ cervical cancer.
* Alcohol or chemical abuse.
* Meningeal carcinomatosis.
* Chemotherapy, radiation therapy, or other anti-tumor therapy during the last four weeks.
* Prior biologic response modifier therapy.
* Refusal in fertile men or women to use effective birth control measures during and for six months after the completion of treatment on study.
* Immune deficiency syndromes, including the following: rheumatoid arthritis, systemic lupus erythematosus, Sjogren's disease, sarcoidosis, vasculitis, polymyositis, glomerulonephritis.
* Compromised lung function:

  * FeV1 < 30% of the predicted value, or
  * DLCO < 30% of the predicted value, or
  * PCO2 > 45 mmHg.
* Any patient enrolled on study whose respiratory symptoms have experienced marked deterioration not related to a known cause, such as pneumonia, congestive heart failure, or pulmonary embolism, will have a repeat PFT evaluation, and if the above parameter values for FeV1, DLCO, or PCO2 are seen, will be excluded from further treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety | 6, 12, 18, 24, and 36 months post enrollment

SECONDARY OUTCOMES:
Immunologic response: CD8, CD4 and NK response | Baseline, Day 1 Week1, Day 1 Week 13, Day 1 Week 19

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Raez, MD, FACP, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Background] Raez LE, Cassileth PA, Schlesselman JJ, Sridhar K, Padmanabhan S, Fisher EZ, Baldie PA, Podack ER. Allogeneic vaccination with a B7.1 HLA-A gene-modified adenocarcinoma cell line in patients with advanced non-small-cell lung cancer. J Clin Oncol. 2004 Jul 15;22(14):2800-7. doi: 10.1200/JCO.2004.10.197. PMID 15254047
- [Result] Raez LE, Podack ER, CD8 T cell response in a phase I study of therapeutic vaccination of advanced NSCLC with allogeneic tumor cells secreting endoplasmic reticulum-chaperone gp96-Ig-peptide complexes. Advances in Lung Cancer 2(1): 9-18, 2013 doi:10.4236/alc.2013.21002